CLINICAL TRIAL: NCT00308893
Title: Brain Derived Neurotrophic Factor (BDNF) Gene Polymorphism and Response to Antidepressants Treatment in Major Depression
Brief Title: BDNF Gene Polymorphism and Antidepressants Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOHP05-WEH/BDNF
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Antidepressants; escitalopram; Genetic polymorphism
MeSH Terms: conditions — Depression | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Treatment response after 3 and 6 weeks
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — Compare BDNF polymorphism among responders and non-responders

SUMMARY:
The main hypothesis is that the therapeutic response and pharmacological resistance to ADs in depressed patients can be associated with a polymorphism for the BDNF gene. The research of allelic forms associated to lesser efficiency or inefficiency of ADs could add to the body of evidence that BDNF mediates the mechanism of action of ADs, and could have important practical implications. We propose to compare in a group of patients with major depression, the allelic variability of the BDNF gene between responders and non-responders after a 3-week period and a 6-week period of SSRI treatment.

DETAILED DESCRIPTION:
* The main objective is to research an association between polymorphism for the BDNF gene and the 3-week and 6-week response to a SSRI treatment (escitalopram) in major depression.
* A case control pilot study without any direct individual benefit (200 patients).
* Study period: 24 months.
* Scores from reliable and validated psychometric scales (Montgomery and Asberg Depression Scale, Mini International Neuropsychiatric Interview) specifically analysing depression dimension at the time of inclusion, after three and six weeks of antidepressant treatment.
* Genetic analysis researching a polymorphism of the BDNF gene is done by a blood sample at the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering a severe depressive episode (according to DSM-IV), evolving since at least 2 weeks before entering the study
* Age superior to 18 years
* Caucasian type
* In absence of any medicinal treatment that could enhance depression: methyldopa, beta-blockers, reserpine,
* In absence of hypothyroidia or anaemia
* Without comorbidity that could affect therapy response : e.g. food disorder, substance abuse or dependence syndrome

Exclusion Criteria:

- Will be excluded from the study the patients for which a modification of the depression diagnosis (according to the DSM-IV criteria) takes place during the period of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2006-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Score on Montgomery and Asberg Depression Rating Scale (MADRS) | At 3 weeks and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wissam EL HAGE, MD, PhD, Principal Investigator — UNIVERSITY HOSPITAL OF TOURS
Locations (1):
- CPU CHRU de Tours, Tours, France

REFERENCES:
- [Result] El-Hage W, Vourc'h P, Gaillard P, Leger J, Belzung C, Ibarguen-Vargas Y, Andres CR, Camus V. The BDNF Val(66)Met polymorphism is associated with escitalopram response in depressed patients. Psychopharmacology (Berl). 2015 Feb;232(3):575-81. doi: 10.1007/s00213-014-3694-z. Epub 2014 Jul 31. PMID 25074447